CLINICAL TRIAL: NCT01139190
Title: A Phase 2 Clinical Trial Evaluating the Incidence of Upper Gastrointestinal Mucosal Damage Following Administration of Either PL3100 or Naproxen in Subjects Who Are at Risk for Developing NSAID-Associated GI Damage
Brief Title: Clinical Trial Evaluating Gastrointestinal Damage Following Administration PL3100 or Naproxen in At-Risk Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PLx Pharma (Industry)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PL-NAP-002; 1RC3AR059535-01 (NIH)
Record Dates: First submitted 2010-06-04; First posted 2010-06-08 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Gastroduodenal Ulcerations; Erosion
Keywords: NSAID-induced gastroduodenal ulcerations or erosion
MeSH Terms: interventions — Naproxen

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PL3100 (Experimental)
  Interventions: Drug: PL3100
- Naproxen (Active Comparator)
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: PL3100 — Oral administration
  Arms: PL3100
Drug: Naproxen — Oral administration
  Arms: Naproxen

SUMMARY:
The purpose of this study is to determine the subchronic gastrointestinal (GI) safety of PL3100 versus Naproxen in normal healthy volunteers.

ELIGIBILITY:
Inclusion Criteria (Selected)

* Male and female healthy adult subjects

Exclusion Criteria (Selected)

* Subject has protocol specified significant medical history.
* Subject is currently participating, or has participated within 30 days prior to study entry, in an investigational drug study.
* Subject has hypersensitivity or contraindications to naproxen, ibuprofen, or other NSAID.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dallas VA Medical Center, Dallas, Texas
  - Houston Center For Clinical Research, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment initiated: 01 July 2010, Multicenter trial: Private practice setting and Veterans Administration gastroenterology clinic.
Pre-assignment Details: No run-in period; subjects screened and enrolled based on review and confirmation of eligibility per inclusion/exclusion criteria. Wash-out period for NSAIDs and gastroprotective agents.
Groups:
- PL3100: Subjects were to take 500 mg of PL3100 (two 250 mg capsules) of study drug twice a day for a total duration of 14.5 days.
- Naproxen: Subjects were to take 500 mg of Naproxen (two 250 mg tablets) of study drug twice a day for a total duration of 14.5 days.
Period: Overall Study
Arm/Group | PL3100 | Naproxen
Started | 38 | 39
Completed | 38 | 38
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PL3100 | Naproxen | Total
Number analyzed (Participants) | 38 | 39 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (5.97) | 55.6 (4.56) | 56.1 (5.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 16 | 19 | 35

OUTCOME MEASURES:

1. Primary Outcome: Degree of GI Injury at Day 15
Description: Degree of mucosal injury was assessed by endoscopy, with the following scoring system:
  Score 0: No Injury Score 1: 1 to 10 petechiae Score 2: > 10 petechiae or 1 to 5 erosions Score 3: 6 to 10 erosions Score 4: > 10 erosions and/or an ulcer
Time Frame: 15 days
Population: Per Protocol Population: subset of participants who had an endoscopy performed at Day 15 reviewed by both blinded endoscopists, was at least 85% compliant with taking the study drug (based on pill counts), who took the final dose drug on the day of the second endoscopy, and who had no other protocol violations that would affect assessments.
Measure: Number; unit: participants
Arm/Group | PL3100 | Naproxen
Number analyzed (Participants) | 34 | 33
participants
  Gastroduodenal Score of 3 or Higher | 23 | 20
  Gastroduodenal Score of 2 or Less | 11 | 13

ADVERSE EVENTS:
Description: Safety Population: all subjects who received at least 1 dose of study drug (naproxen or PL3100) under the study protocol.
Arm/Group | PL3100 | Naproxen
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/39
Other Adverse Events (participants affected / at risk) | 23/38 | 7/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PL3100 (N=38) | Naproxen (N=39)
Abdominal Cramps (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 1 (1)
Nasusea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Stomach ulcer (Gastrointestinal disorders) | 7 (7) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less